CLINICAL TRIAL: NCT05934513
Title: A Phase Ib/II, Multicentre, Open-label Study to Assess the Efficacy, Safety/ Tolerability and Pharmacokinetic of GFH009 Monotherapy in Patients with Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Brief Title: A Study of GFH009 Monotherapy in Patients with Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFH009X1201
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-09

CONDITIONS: Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GFH009 (Experimental): all patients will be administrated with GFH009
  Interventions: Drug: GFH009

INTERVENTIONS:
Drug: GFH009 — patients are planned to be administrated with GFH009 every week in a 21 days cycle, intravenous infusion

SUMMARY:
This is a multicentre, open-label phase Ib/II study. The purpose of the study is to assess the efficacy, safety/ tolerability and pharmacokinetic of GFH009 monotherapy in patients with relapsed or refractory peripheral T-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years and ≤ 75 years.
2. Written informed consent must be obtained prior to any screening procedures.
3. Patients with histologically confirmed relapsed or refractory peripheral T-cell Lymphoma.
4. Must have received and failed at least 2 but no more than 5 prior lines of therapies .
5. Presence of at least 1 radiographically measurable lymphoma disease lesion (according to the Lugano criteria).
6. Fresh tumor tissue or archival tumor tissue must be confirmed to be available at screening.
7. Eastern Cooperative Oncology Group performance status of ≤ 2.
8. Adequate haematologic and organ function at screening.
9. Life expectancy ≥ 12 week.
10. Recovery to grade 0-1 from adverse events related to prior anti-tumor therapy except alopecia, fatigue and < Grade 2 sensory neuropathy.
11. For women of childbearing potential, she must consent to use highly effective methods of contraception during GFH009 treatment and for an additional 90 days after the last administration of study drug. Men with a partner of childbearing potential, must consent to use highly effective methods of contraception during GFH009 treatment and for an additional 90 days after the last administration of study drug

Exclusion Criteria:

1. Diagnosis of Cutaneous T-cell lymphoma .
2. Symptomatic central nervous system (CNS) metastases, leptomeningeal disease, or spinal cord compression.
3. Patients with severe hemophagocytic syndrome at screening.
4. Presence of uncontrolled third space effusion
5. Patients who have received chemotherapy, radiotherapy or anti-tumor Chinese traditional medicines within 2 weeks prior to starting study drug; or undergone major surgery with 4 weeks; or received targeted therapy within 4 weeks or 5 half-lives whichever is shorter; or received immunotherapy.
6. History of allogeneic stem cell transplant or autologous HCT within 90 days before screening.
7. Attend other clinical trial within 2 weeks prior to starting study drug.
8. History of previous exposure to any other CDK9 inhibitor.
9. Concurrent malignancy within 5 years prior to entry
10. Uncontrolled pulmonary fibrosis, active lung diseases or interstitial lung disease.
11. Severe cardiovascular disease
12. Subjects with high risk of gastrointestinal hemorrhage.
13. Uncontrolled infective diseases.
14. Ongoing therapy with corticosteroids greater than 20 mg of prednisone or its equivalent per day and the duration of treatment was more than 14 days.
15. Concomitant medications that are strong CYP3A4 inhibitors or strong inducers within 7 days prior to the first dose. Avoid consumption of Seville orange (and juice), grapefruit or grapefruit juice, grapefruit hybrids, pomelos, star citrus fruits or St. John's wort within 7 days of first dose.
16. Major surgery within 4 weeks prior to study entry or surgery is under schedule in the short run.
17. Pregnant or breast-feeding female.
18. Any uncontrolled intercurrent illness or condition that in the judgement of the investigator may endanger the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: adverse events | From Screening (Day -28 to Day-1) until disease progression or survival until death (approximately 6 months)
  Incidence of intolerable toxic events, incidence and severity of adverse events (AEs) and serious adverse events (SAEs)
Phase II: Objective Response Rate | From Screening (Day -28 to Day-1) until disease progression or survival until death (approximately 6 months)
  ORR(Objective Response Rate)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No